CLINICAL TRIAL: NCT05013255
Title: Pioglitazone Therapy Targeting Fatigue in Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Jessica Partin, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2103254164
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Muscle Fatigue
MeSH Terms: conditions — Breast Neoplasms | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pioglitazone 15mg Dose (Active Comparator): Subjects will be given PIO 15mg once daily, based on the randomization lists prepared by the WVUCI Biostatistics Core. This is a 1:1:1 randomization (10 in each group) without any planned stratification.
  Interventions: Drug: Pioglitazone 15mg
- Pioglitazone 30mg Dose (Active Comparator): Subjects will be given PIO 30mg once daily, based on the randomization lists prepared by the WVUCI Biostatistics Core. This is a 1:1:1 randomization (10 in each group) without any planned stratification.
  Interventions: Drug: Pioglitazone 30 mg
- No Drug (No Intervention): Subjects will be assigned to a no drug control group based on the randomization lists prepared by the WVUCI Biostatistics Core. This is a 1:1:1 randomization (10 in each group) without any planned stratification.

INTERVENTIONS:
Drug: Pioglitazone 15mg — PIO 15mg orally once daily for 2 weeks
  Other Names: Actos
  Arms: Pioglitazone 15mg Dose
Drug: Pioglitazone 30 mg — PIO 30mg orally once daily for 2 weeks
  Other Names: Actos
  Arms: Pioglitazone 30mg Dose

SUMMARY:
The goal of this project is to evaluate the therapeutic potential of pioglitazone (PIO) to target underlying mechanisms that promote muscle fatigue in patients with breast cancer. This represents an off-label use of this compound, both in terms of the patient population and the clinical phenotype targeted. The central research hypothesis of this study is that daily pioglitazone will restore transcriptional downregulation of pathways within skeletal that promote fatigue.

DETAILED DESCRIPTION:
Fatigue is commonly reported in cancer patients, but is not treated due to the absence of viable therapies. At the time of diagnosis, prior to treatment, nearly all breast cancer patients have some degree of muscle dysfunction resulting in fatigue that ranges from mild to debilitating and may worsen with chemotherapy, radiation, and/or surgery. A significant gap in knowledge exists with respect to targetable mechanisms to alleviate fatigue in patients with cancer. The goal of this project is to evaluate the therapeutic potential of pioglitazone (PIO) to target underlying mechanisms that promote muscle fatigue in patients with breast cancer. This represents an off-label use of this compound, both in terms of the patient population and the clinical phenotype targeted. The central research hypothesis of this study is that daily pioglitazone will restore transcriptional downregulation of pathways within skeletal that promote fatigue. The investigators believe this trial will provide the clinical data on optimal PIO dose to affect muscle gene expression in patients with breast cancer. This data will be used to support a larger clinical trial in patients with and without breast cancer to determine PIO therapy effects on muscle fatigue.

Pioglitazone is an FDA-approved drug that is used to treat insulin resistance in patients with diabetes by targeting PPARγ activity, although this drug also affects mitochondrial function through PPARγ regulation. Therefore, the investigators will test the central research hypothesis that daily pioglitazone will restore transcriptional downregulation of pathways within skeletal that promote fatigue. Specific Aim 1 will determine the molecular signature within skeletal muscle in response to low dose and high dose pioglitazone therapy. It is predicted that daily pioglitazone therapy will reverse the breast cancer-associated downregulation of mitochondrial and metabolic genes in skeletal muscle. Specific Aim 2 will determine the effects of low dose and high dose pioglitazone therapy on perceptions of fatigue. It is predicted that daily pioglitazone therapy will improve patient reported perceptions of fatigue.

This is a Phase 2B Trial to determine the lowest effective dose of pioglitazone for affecting skeletal muscle gene expression in breast cancer patients without diabetes (dose-finding study). At the time of registration, subjects will be randomized to either the low dose (15mg PIO; n=10) or the high dose (30mg PIO; n=10) group, or a no-drug control group (n=10). Drug therapy will last for 2 weeks, leading into a scheduled mastectomy. Subjects will be provided with a 2 week supply of PIO on Study Day 1 to be taken orally once per day. Following surgery and muscle biopsy collection subjects will be followed for adverse events, fatigue and body composition for 30 days through their first post-op visit. The total study duration will be 6-weeks (2 weeks of drug treatment + 4 weeks until follow-up visit).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed luminal (ER+/PR+ Her2/neu-) Breast Cancer.
* Subjects must have received no prior therapies besides chemotherapy in the neoadjuvant setting.
* Subject must have a planned surgical (mastectomy) date within 2 weeks of starting treatment.
* 5 Subjects must have normal organ as defined below:

  * Hemoglobin within normal institutional limits (or >10?)
  * Fasting Blood Glucose within normal institutional limits
  * Serum Creatinine within normal institutional limits
  * Liver Function (AST and ALT, Alk phosphatase, Total Bilirubin) within normal limits
* Subject does not have a prior diagnosis of diabetes or currently taking any medications to lower blood glucose levels.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior diagnosis of Congestive Heart Failure (CHF), Bladder cancer, osteoporosis, bariatric surgery
* Subjects receiving any other investigational agents or known agents to have a major interaction with PIO to include clopidogrel, gatifloxacin, gemfibrozil, leflunomide, lomitapide, lumateperone, mipomersen, pexideartinib and teriflunomide, insulin, Lyrica, Synthroid.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pioglitazone.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, active alcoholism or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding are excluded from this study because Pioglitazone has the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with PIO, breastfeeding should be discontinued if the mother is treated with PIO. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Gene Expression | Up to 6 weeks
  evaluate the ability of daily pioglitazone therapy to attenuate the transcriptional downregulation of a gene network within skeletal muscle that is integral to mitochondrial bioenergetics, with PPARγ central to this network. The outcome measure will be RNA-Sequencing and gene expression analysis from muscle biopsies obtained from subjects following either low dose or high dose pioglitazone therapy.

SECONDARY OUTCOMES:
Muscle Fatigue | Up to 6 weeks
  Assess the fatigue in subjects with breast cancer that are being treated with pioglitazone, as measured by the FACT-F questionnaire. 5 point Likert-type scale where 0= Not at all, 1= A little bit, 2= Somewhat, 3= Quite a bit, 4= Very much.
Body Weight | 2 weeks
  Monitor body weight for loss or gains in subjects receiving low dose and high dose pioglitazone for 2 weeks prior to a scheduled mastectomy

CONTACTS AND LOCATIONS:
Overall Officials: Kristin H Lupinacci, DO, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Cancer Institute, Morgantown, West Virginia, United States